CLINICAL TRIAL: NCT02637414
Title: Flourishing App: Evaluation of the Effectiveness of a Well-being Application for Mobile Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Principal Investigator, Elisa Kozasa, PhD, Hospital Israelita Albert Einstein
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HIAE_App Florescer
Record Dates: First submitted 2015-12-11; First posted 2015-12-22 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Emotional Stress
Keywords: Stress; Well-being; Positive psychology
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control App (No Intervention): Initially this control group will have access to a Control App and after 8 weeks this goup will receive the intervention (Flourishing App Program).
- Flourishing App Program (Experimental): This group will receive the intervention Flourishing App Program and after that it will not receive any other intervention.
  Interventions: Behavioral: Flourishing App Program

INTERVENTIONS:
Behavioral: Flourishing App Program — This intervention is based on relaxation, well-being promotion, meditation practices and positive psychology principles. The program is being evaluated in a classroom format into another project and was adapted for this project in the application format for mobile devices. It will last for 8 weeks, with trainings of 15 to 25 minutes, four times a week.
  Arms: Flourishing App Program

SUMMARY:
This protocol proposes a well-being program, delivered through an application for mobile devices, based on meditation and positive psychology principles such as human development, the improvement of virtues, quality of life and well-being. The investigators hypothesize that this program offered in mobile application may promote well-being and reduce stress related problems in the participants.

Objectives: To evaluate the effectiveness of a well-being program delivered through an application for mobile devices in a sample of employees who work in a company (Natura Inovação/Cosméticos) and in a hospital (Hospital Israelita Albert Einstein).

Methods: Two hundred and fifty employees from Natura Inovação/Cosméticos and 250 employees from Hospital Israelita Albert Einstein will be recruited. The participants will be randomized in two groups of 125 participants each one, half of them in the control group (GC) and the other half to the intervention group (GI), by institution.

DETAILED DESCRIPTION:
Introduction: Stress related disorders may result in absenteeism and less productivity in companies. This protocol proposes a well-being program, delivered through an application for mobile devices, based on meditation and positive psychology principles such as human development, the improvement of virtues, quality of life and well-being. In the modern world not all people are willing to attend classroom training for several reasons. In this sense, the investigators hypothesize that this program offered in mobile application may promote well-being and reduce stress related problems in the participants.

Objectives: To evaluate the effectiveness of a well-being program delivered through an application for mobile devices in a sample of employees who work in a company (Natura Inovação/Cosméticos) and in a hospital (Hospital Israelita Albert Einstein).

Methods: Two hundred and fifty employees from Natura Inovação/Cosméticos and 250 employees from Hospital Israelita Albert Einstein will be recruited. The participants will be randomized in two groups of 125 participants each one, half of them in the control group (GC) and the other half to the intervention group (GI), by institution. The GI will participate in the Flourishing App Program, for eight weeks, while the GC will have access to a Control App. Then, after the evaluations, the GC will receive the intervention (Flourishing App Program), while the first group will not receive any intervention. Questions will be applied to evaluate the levels of stress and well-being of participants before and after the program and before and after each training period.

ELIGIBILITY:
Inclusion Criteria:

* Female aging from 18 to 60
* Complete higher education
* Employees from Natura Inovação/Cosméticos and from Hospital Israelita Albert Einstein

Exclusion Criteria:

* none

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Actual)
Dates: Start 2016-01; Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Changes in subjective symptoms of well-being at work | baseline, 4 weeks, 8 weeks
  Sliding scale for stress level from 0 to 100
Changes in subjective symptoms of stress | baseline, 4 weeks, 8 weeks
  Sliding scale for well-being level from 0 to 100

SECONDARY OUTCOMES:
Changes in subjective symptoms of stress at the moment assessed using the sliding scale for stress | four times a week, before and after the period of each class (20 min)
  Sliding scale for stress level from 0 to 100
Changes in subjective symptoms of well-being at the moment assessed using the sliding scale for well-being | four times a week, before and after the period of each class (20 min)
  Sliding scale for well-being level from 0 to 100

CONTACTS AND LOCATIONS:
Overall Officials: Elisa H Kozasa, PhD, Principal Investigator — Instituto do Cérebro- Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, Brazil

REFERENCES:
- [Derived] Coelhoso CC, Tobo PR, Lacerda SS, Lima AH, Barrichello CRC, Amaro E Jr, Kozasa EH. A New Mental Health Mobile App for Well-Being and Stress Reduction in Working Women: Randomized Controlled Trial. J Med Internet Res. 2019 Nov 7;21(11):e14269. doi: 10.2196/14269. PMID 31697244